CLINICAL TRIAL: NCT03756116
Title: Effect of Papillary Epinephrine Spraying for the Prevention of Post-ERCP Pancreatitis in Patients Received Sublingual Nitroglycerin: A Multi-center, Single-blind, Randomized Controlled Trial
Brief Title: Effect of Papillary Epinephrine Spraying for the Prevention of Post-ERCP Pancreatitis in Patients Received Octreotide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEP-17-07
Record Dates: First submitted 2018-10-16; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-10

CONDITIONS: Post-ERCP Acute Pancreatitis; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epinephrine sprayed on the papilla (Experimental): Patients received sublingual Nitroglycerin will receive 20 ml of 0.02% epinephrine sprayed on the duodenal papilla before the withdrawal of endoscope.
  Interventions: Procedure: Epinephrine sprayed on the papilla
- Saline sprayed on the papilla (Active Comparator): Patients received sublingual Nitroglycerin will receive 20 ml of normal saline sprayed on the duodenal papilla before the withdrawal of endoscope; followed by octreotide.
  Interventions: Procedure: Saline sprayed on the papilla

INTERVENTIONS:
Procedure: Epinephrine sprayed on the papilla — Patients received sublingual Nitroglycerin will receive 20 ml of 0.02% epinephrine sprayed on the duodenal papilla before the withdrawal of endoscope.
  Arms: Epinephrine sprayed on the papilla
Procedure: Saline sprayed on the papilla — Patients received sublingual Nitroglycerin will receive 20 ml of normal saline sprayed on the duodenal papilla before the withdrawal of endoscope.
  Arms: Saline sprayed on the papilla

SUMMARY:
Post-endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis (PEP) is the most common complication with high costs, significant morbidity and even mortality. The major mechanisms of PEP is the papillary edema which is caused by manipulations during cannulation or endoscopic treatment. The papillary edema may cause temporary outflow obstruction of pancreatic juice, and then increase ductal pressure, resulting in the occurrence of pancreatitis. Nitroglycerin can reduce the Oddis sphincter tension, the internal pressure of the biliary tract and the pancreatic duct. Therefore, it is widely used in clinical to prevent and treat pancreatitis. Many studies found nitroglycerin might be effective in preventing PEP. And topical application of epinephrine on the papilla may reduce papillary edema by decreasing capillary permeability or by relaxing the sphincter of Oddi. There are reports that epinephrine sprayed on the papilla may be effective to prevent PEP.

The investigators therefore designed a prospective randomized trial to determine whether routine using papillary epinephrine spraying in patients received octreotide can reduce post-ERCP pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. ERCP surgery is required
2. Signed inform consent form and agreed to follow-up on time.

Exclusion Criteria:

1. Acute pancreatitis.
2. Pregnancy or history of allergy to epinephrine.
3. Serious liver, kidney, heart and coagulation disorders
4. Unwilling or inability to provide consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-ERCP pancreatitis in the groups | 48 hours after ERCP
  The primary outcome is the incidence of PEP as defined by the consensus guidelines as 1) New or increased abdominal pain that is clinically consistent with a syndrome of acute pancreatitis without other acute abdominal diseases,such as gastrointestinal perforation,acute cholecystitia and acute cholangitis and etc, and 2) amylase or lipase ≥ 3x the upper limit of normal 48 hours after the procedure.

SECONDARY OUTCOMES:
Others complications | 1 weeks after ERCP
  Others complications are the cute cholecystitia, acute cholangitis,hemorrhage and perforation，et al.

CONTACTS AND LOCATIONS:
Overall Officials: Miao Lin, Principal Investigator — Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China